CLINICAL TRIAL: NCT02641665
Title: Measurement of Four Plasma Biomarkers for Risk Stratification and Determination of Functional Recovery After Cardiac Valve Surgery
Brief Title: Plasma Biomarkers in Cardiac Valve Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor, Head of Department, University of Liege
Other Study IDs: 2016001
Record Dates: First submitted 2015-12-22; First posted 2015-12-29 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Elective Valvular Cardiac Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Arterial blood
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Cardiac valve surgery — Aortic or mitral valve replacement/repair performed in isolation of in addition to coronary artery bypass graft(s).

SUMMARY:
The level of four biomarkers will be measured in the patients' plasma after induction of anaesthesia. There biomarkers are NT-ProBNP, ST2, Galectin-3 and GDF-15. The level of these marker will then be correlated with early (30 days) and late (one year) patients' prognosis and with functional recovery (MLHFQ score).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Elective/urgent aortic or mitral valve surgery in isolation or combined with CABG

Exclusion Criteria:

* Emergency or salvage surgery
* Inability to consent
* Previous cardiac surgery
* Stage IV or V CDK (GFR ≤ 30 ml/min) or dialysis
* Active Endocarditis
* Liver cirrhosis
* Chronic atrial fibrillation
* Pacemaker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing elective or urgent cardiac valve surgery in isolation of in combination with CABG.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2016-01; Primary Completion 2017-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Composite primary outcome | 30 days
  In hospital or 30-days mortality or inotropic support during more than 48 hours or lengthy of ICU stay longer than 5 days

SECONDARY OUTCOMES:
ICU readmission | 30 days
Post-operative AKI | 48 hours
  AKIN stage during the first 48 hours
Ejection fraction | 1 year
  EF at 30 days and at 1 year
NYHA | 1 year
  NYHA class at 30 days and at 1 year
MLHFQ | 1 year
  Minnesota living with heart failure questionnaire at 30 days and at 1 year
reshopitalisation | 1 year
  hospital admission for cardiac failure during the first postoperative year
one year mortality | 1 year
  mortality during the first postoperative year.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU of Liege, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No